CLINICAL TRIAL: NCT04580368
Title: Testing Drug Efficacy in Cystic Fibrosis Through N-of-1 Trials
Acronym: Nof1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N of 1_2019-0545
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: CFTR modulators; cystic fibrosis; HNE; human nasal epithelial cells; NPD; nasal potential difference; air-liquid interface; N-of-1
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: N of 1 trial using an individual patient as their own control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CFTR modulator or other therapies (Experimental): CFTR modulator or active therapy
  Interventions: Drug: CFTR Modulators

INTERVENTIONS:
Drug: CFTR Modulators — Participants with rare mutations will receive active therapy in N-of-1 design with participants serving as their own control

SUMMARY:
The purpose of this study is to validate and utilize a personalized medicine approach to identify potential treatments with current FDA approved CFTR modifiers for non-approved CF gene mutations. The study will perform ex vivo testing of CFTR function and current marketed CFTR modulating drugs on expanded nasal cells at Cincinnati Children's Human Nasal Epithelium (HNE) Core Laboratory. The results will be confirmed and translated into bedside care through an N of 1 trial to determine effectiveness of treatment.

DETAILED DESCRIPTION:
This is a protocol for the development of personalized treatments from bench to bedside for rare CF mutations. The protocol will start with the current FDA-approved CFTR modulators and continue to add newly developed CF drug therapies to the potential treatment testing options as they are approved for market. This is a single-center study enrolling subjects with rare CFTR variants who are prescribed CFTR modulators by their treating physician. This decision may be based on the patient's genotype (e.g., a patient with a CFTR mutation known to respond to drug) or based on preclinical HNE model testing; regardless, the decision to start a modulator is made by the subject's physician, not by the study team.

The N-of-1 design includes a basic research component using nasal brushings which will be expanded in the HNE Core Lab and tested with CFTR modulating drug therapies. Based on the HNE culture's reactivity to the tested CFTR modulating drugs, an N-of-1 trial will be initiated to test if this translates to therapeutic benefit.

The CFTR modulating drugs that are currently FDA approved and will be tested in this study include ivacaftor and the combination drugs orkambi (ivacaftor/lumacaftor), symdeko (ivacaftor/tezacaftor), and trikafta (elexacaftor/tezacaftor/ivacaftor). All will be used in clinically prescribed dosages and within the FDA approved age ranges.

For HNE testing, subjects will fall into two pools. The first will have already undergone HNE model testing with positive results. These subjects will proceed directly to N-of-1 testing without additional ex vivo studies. The second group will have been referred for N-of-1 testing based on their CFTR genotype, having not previously undergone HNE testing. This group will have HNEs harvested at the initial visit, and HNE testing will occur in parallel to N-of-1 testing.

For the N-of-1 portion of this trial, subjects will undergo a 14-day run-in period, followed by an observational 28-day block of non-treatment. This will be followed with a 14-day washout period, and then by a 28-day block of modulator treatment, with a final 14-day washout period and a 14-day follow-up period before study completion. Repeated assessments will occur at the beginning and end of each 28-day block. Participants will therefore be on study for approximately 112 days. This protocol will remain open indefinitely to develop treatment options for patients with new and not well defined forms of Cystic Fibrosis and CFTR disorders.

At this time, CFTR modulator drugs can only be filled in specialty pharmacies, and is not on formulary at CCHMC. While the development of a specialty pharmacy was in process at CCHMC, this progress has halted due to the COVID-19 pandemic. Because the drugs cannot be filled internally, the Investigational Drug Service is unable to dispense them or provide placebo for blinded studies. Because understanding the individual response to these compounds and the relationship of that response to HNE models is critical, this study will move forward in an open-label fashion. If the CCHMC specialty pharmacy is successfully opened, we anticipate a revision to modify this protocol to a double-blinded, placebo-controlled crossover, however, this is not currently possible. This change has been discussed with the funding agency (NIH / NIDDK), who are in agreement.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (and assent when applicable)
* Willing and able to adhere to the study visit schedule and protocol requirements
* Male or Female ≥6 years old and within the FDA-approved range for the proposed modulator drug

  * Ivacaftor: ≥4 months old
  * Lumacaftor/Ivacaftor: 2 years old
  * Tezacaftor/Ivacaftor: 12 years old
  * Elexacaftor/Tezacaftor/Ivacaftor: ≥12 years old
* At least one rare CFTR variant (incidence of <5% of the CF population)
* Documentation of a CF diagnosis as evidenced by one or more clinical features of CF plus at least one of the following:

  * Sweat Chloride ≥60mmol/L by quantitative pilocarpine iontophoresis
  * Two mutations in the CFTR gene
  * Abnormal nasal potential difference (NPD) testing supportive of a CF diagnosis
* FEV1 > 50% predicted for age
* Stable chronic CF therapies with no changes in >28 days (except for chronic cycled inhaled antibiotics such as tobramycin)
* Prescribed CFTR modulator by a licensed physician
* No contraindication to treatment with the selected drug at the time of treatment initiation

Exclusion Criteria:

* Presence of any condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the patient and/or quality of the data
* For women of child bearing potential:

  * Positive pregnancy test or known pregnancy at Visit 1
  * Lactating
  * Unwilling to practice a medically acceptable form of contraception (acceptable forms include abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent), unless surgically sterilized or postmenopausal during the study
* BMI < 10th percentile for age (if <18 years old) or < 20kg/m2 (if ≥18 years old)
* FEV1 ≤ 50% predicted for age
* Growth of CF pathogens from sputum cultures that are associated with unstable disease (e.g., nontuberculous mycobacteria, Burkholderia spp) within six months of enrollment
* Concomitant use of CYP3A inducers or inhibitors (e.g., voriconazole, fluconazole, rifampin) or prednisone (>20mg daily)
* Concomitant conditions:

  * Poorly controlled diabetes mellitus (HbA1c >8.5 or glucosuria as noted below)
  * Advanced CF liver disease (cirrhosis with portal hypertension, ascites, or abnormal liver laboratory testing as noted below)
  * End stage renal disease
  * History of organ transplantation
  * Additional medical conditions that in the opinion of the Investigator place the patient at risk of participation or may impact the patient's ability to complete the trial (e.g., uncontrolled depression, anxiety disorder, poor adherence to CF therapies, active ABPA)
* Any of the following abnormal laboratory values at the Screening Visit:

  * CBC
  * WBC >15,000 K/mcL or ANC <1,500 K/mcL
  * Hemoglobin <10 gm/dL
  * Platelets <50,000 K/mcL
  * Chemistries
  * >2+ Glucosuria
  * Clinically significant abnormalities as assessed by the Investigator
  * Glomerular filtration rate ≤50 mL/min/1.73 m2 (calculated by the Counahan-Barratt equation)
  * Hepatic Function Testing / Coagulation Testing
  * ≥3 × upper limit of normal (ULN) aspartate aminotransferase (AST)
  * ≥3 × ULN alanine aminotransferase (ALT)
  * ≥3 × ULN gamma-glutamyl transpeptidase
  * Total or direct bilirubin >2 × ULN
  * INR > 1.5 x ULN
  * Positive pregnancy test

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
ppFEV1 | 16 weeks
  Absolute change in ppFEV1 of 5% or greater

CONTACTS AND LOCATIONS:
Locations (1):
- CCHMC, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No